CLINICAL TRIAL: NCT06381791
Title: Cannabidiol (CBD) As A Pain Adjunct in Orthopedic Surgical Patients: A Randomized Control Trial
Brief Title: CBD for Pain Following Orthopedic Shoulder Surgery
Acronym: CBD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, The John S. Dunn Chair in Orthopedic Surgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00036811
Record Dates: First submitted 2024-04-11; First posted 2024-04-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Shoulder Osteoarthritis; Rotator Cuff Injuries
Keywords: CBD; Cannabidiol; Epidiolex
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, double-blinded controlled trial. Patients will be recruited in clinic preoperatively prior to their scheduled procedure. Patients and the treating physician/research study team will be blinded to the treatment arm. Patients will be randomized to either the test group, which will be prescribed Epidiolex (cannabidiol) postoperatively in addition to the standard pain regimen, or the control group, which will have a placebo provided in addition to the standard pain regimen.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epidiolex (cannabidiol) (Experimental): Patients randomized to the Epidiolex group will take 150mg of Epidiolex with food twice daily for 14 days beginning the day of surgery.
  Interventions: Drug: Epidiolex
- Placebo (Placebo Comparator): Patients randomized to the placebo group will take 150mg of oral placebo solution with food for 14 days beginning the day of surgery.
  Interventions: Drug: Placebo oral solution

INTERVENTIONS:
Drug: Epidiolex — 150mg of Epidiolex
  Other Names: Cannabidiol Oral Solution
  Arms: Epidiolex (cannabidiol)
Drug: Placebo oral solution — 150mg of Placebo oral solution
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of the study is to learn if Epidiolex (cannabidiol) works as a additional pain medication in patients who have had orthopedic shoulder surgery. It is also to learn about safe dosages and identify any side effects after surgery.

Researchers will compare Epidiolex to a placebo solution to see if Epidiolex lowers pain after shoulder surgery.

Participants will:

* track their pain and what medications they use every day in a provided pain diary. A researchers will call every seven days to check on the participant and diary.
* Complete two short surveys. Once before surgery and once after.
* Have bloodwork tested after surgery

DETAILED DESCRIPTION:
Subjects will be randomized according to their surgery type. They will receive either the Epidiolex cannabidiol in addition to their standard of care pain regimen or a placebo in addition to their standard of care pain regimen. They will be asked to track a pain diary for 2 weeks postoperatively.

A member of the research team will conduct a follow-up telephone call on day 7 to assess subjects' drug compliance. Subjects will also be contacted for a safety monitoring call at day 7 and 1 week after completion of treatment in which they will disclose type, severity, onset, and duration of any adverse events. In addition, they will complete a suicidal assessment10 See attached safety screening document. After the 2 weeks, subjects will return the pain diary and vial of CBD/placebo at their postoperative appointment.

Subjects will also be asked to complete validated questionnaires via Houston Methodist's Redcap system once before surgery and again at 14 days postop. The surveys are with regards to sleep, activity, and pain and should take no more than 15 minutes to complete.

At their standard of care postoperative visit (11-17 days following surgery), another liver panel will be taken and their final safety monitoring screening will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing one of the following orthopedic shoulder surgeries:

  * Total shoulder arthroplasty
  * Reverse total shoulder arthroplasty
  * Shoulder hemiarthroplasty
  * Rotator cuff repair
* Receiving standard anesthesia during surgery
* If a subject is of reproductive potential, they must be on effective contraception one month prior, during treatment, and one month following treatment.

Exclusion Criteria:

* Not above the age of 18 years old
* History of revision shoulder arthroplasty
* History of liver disease or impairment
* Are currently taking valproate or clobazam
* Are currently taking a moderate/strong CYP3A4 or CYP2C19 inhibitor
* Are currently taking a strong CYP3A4 or CYP2C19 inducer
* Are currently taking narcotics
* History of substance/alcohol abuse
* Those currently or previously under the care of a pain management specialist
* History of marijuana/cannabidiol (not including topical) regular use within the past 6 months
* Allergy related to cannabidiol
* Allergy related to sesame seeds
* Pregnancy (As part of standard of care, all female participants will be administered a urine pregnancy test prior to surgery. A negative test result is required to participate in the study.)
* If you are taking any medications with known risks for suicidal behavior and ideation
* If you have a diagnosed psychiatric or sleeping disorder
* If you are actively breastfeeding
* Patients currently taking central nervous system (CNS) depressants
* Patients currently taking other drugs with known hepatotoxicity
* Vulnerable populations.

Patients taking concomitant medications which are substrate of uridine 5'-diphospho-glucuronosyltransferase 1-9 (UGT1A9), uridine diphosphate-glucuronosyltransferase 2B7 (UGT2B7), CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, and P-gp will be monitored for potential adverse events based on the Epidiolex® label for the concomitant medication being used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary - Pain Journal | 2 weeks
  Evaluation of postoperative pain journal responses from subjects. The pain diary will track their pain level on a Visual Analogue Scale (VAS) and their documented pain medication usage.

SECONDARY OUTCOMES:
Survey Data | 2 weeks
  Evaluation of the survey data and questionnaires from baseline to the end of the two weeks post operative period.
Pain Disability Index (PDI) | 2 weeks
  This survey is designed to measure the degree to which aspects of a participant's life are disrupted by chronic pain. Each item on the survey is rated on an eleven point scale from no disability (0) to worst disability (10).
Pain, Enjoyment, General Activity (PEG) Scale | 2 weeks
  This survey tracks a participant's pain intensity and pain interference. Each item on the survey is rated on an eleven point scale from 0 to 10 with different measures at either end of the scale depending on which item (intensity or interference) is being evaluated.
Patient Health Questionnaire 4 (PHQ-4): The four-item patient health questionnaire for anxiety | 2 weeks
  This survey measures how frequently a patient was bothered by symptoms of anxiety or depression. It is measured on a four point scale from 0-3 with each number corresponding to how often a patient experienced a symptom with 0 being not at all, and 3 being nearly every day.
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks
  This survey assesses the amount and quality of sleep that a patient has experienced in the last month. It is measured both with general free response questions and scaled questions reflecting frequency or lack thereof for a given issue (rated from Not during the past month to Three or more times a week).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No